CLINICAL TRIAL: NCT03635996
Title: Multi-Centre, Open-Label, Safety Study of Etripamil Nasal Spray in Spontaneous Episodes of Paroxysmal Supraventricular Tachycardia The NODE-302 Trial (Extension of NODE-301)
Brief Title: Safety Study of Intranasal Etripamil for the Termination of Spontaneous Episodes of Paroxysmal Supraventricular Tachycardia (PSVT). NODE-302
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was stopped by the Sponsor
Sponsor: Milestone Pharmaceuticals Inc. (Other)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSP-2017-1158
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Results first posted 2023-04-24 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2021-03

CONDITIONS: Paroxysmal Supraventricular Tachycardia
Keywords: Paroxysmal supraventricular tachycardia; cardiac monitoring; atrioventricular nodal reentrant tachycardia; atrioventricular reciprocating tachycardia; calcium channel blocker; conversion rate
MeSH Terms: conditions — Tachycardia, Ventricular; Tachycardia, Atrioventricular Nodal Reentry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Etripamil NS 70 mg (Experimental): The dose of etripamil to be evaluated in NODE-302 is 70 mg.
  Interventions: Drug: Etripamil NS 70 mg; Device: Aptar Pharma Nasal Spray Bidose System

INTERVENTIONS:
Drug: Etripamil NS 70 mg — All patients will receive a total of 200 micro-liters of etripamil NS 70 mg via the Aptar Pharma Nasal Spray Bidose System each time they self-administer study drug.
  Other Names: MSP-2017
Device: Aptar Pharma Nasal Spray Bidose System — Patients will self-administer the study drug using the Aptar Pharma Nasal Spray Bidose System. The devices will be prefilled and packaged into child-resistant boxes.Instructions for its use will be provided in the study drug box.

SUMMARY:
The primary objective of this study is to evaluate the safety of etripamil nasal spray (NS) 70 mg when self-administered by patients with an episode of Paroxysmal Supraventricular Tachycardia in an outpatient setting (i.e., without medical supervision).

DETAILED DESCRIPTION:
The NODE-302 study is an extension of the NODE-301 efficacy study. It is a multi-centre, open label study designed to evaluate the safety of etripamil NS 70 mg when self-administered by patients for spontaneous episodes of PSVT in an outpatient setting. All patients randomized in the NODE-301 study and who meet the inclusion and exclusion criteria of the NODE-302 study are eligible for the NODE-302 study.

After each episode of PSVT, patients will have the option to continue in the NODE-302 study and manage subsequent episodes of PSVT with etripamil NS 70 mg if they do not meet any withdrawal criteria.

Each episode of PSVT will be documented by an ambulatory cardiac monitoring system (CMS) that will be placed on the chest by the patient or caregiver when symptoms begin, and will record at least 5 hours of continuous ECG.

The study will include a Qualification Visit, a Treatment Period(s) , a Follow-up Visit(s) ,a Final Study Visit and if necessary an Early Termination Visit if the patient withdraws from the study after taking etripamil NS 70 mg and had a Follow-up Visit, or the patient withdraws from the study and did not take etripamil NS 70 mg.

ELIGIBILITY:
Inclusion Criteria

Patients who meet all of the following criteria will be eligible to participate in the study:

1. Male or female patients at least 18 years of age;
2. Signed the NODE-302 written informed consent;
3. Previously randomized in the NODE-301 study:

   * Received the study drug to treat symptoms the patient believed were consistent with an episode of PSVT during the NODE-301 study, irrespective of the study drug efficacy; OR
   * Did not experience an episode of PSVT or did not use the study drug at the time of the NODE-301 study completion;
4. Willing and able to comply with all aspects of the study;
5. Females of childbearing potential who are sexually active must agree to use an approved highly effective form of contraception from the time of signed informed consent until 30 days after the last administration of study drug. Females of childbearing potential should have a negative urine pregnancy test result at the Qualification Visit and at the Follow-up Visit(s), and must use an approved form of contraception between the 2 visits. Approved forms of contraception include hormonal intrauterine devices and hormonal contraceptives (oral birth control pills, Depo Provera®, patch, or other injectables) together with supplementary double barrier methods, such as condoms or diaphragms with spermicidal gel or foam;

   The following categories define females who are NOT considered to be of childbearing potential:
   * Premenopausal females with 1 of the following:

     1. Documented hysterectomy,
     2. Documented bilateral salpingectomy, or
     3. Documented bilateral oophorectomy, or
   * Postmenopausal females, defined as having amenorrhea for at least 12 months without an alternative medical cause; and
6. Male patients, except those who are surgically sterile, must use an approved highly effective form of contraception during the 3 days after study drug administration.

Exclusion Criteria

Patients who meet any of the following criteria will be excluded from participation in the study, including but not limited to:

1. Evidence of new severe arrhythmia discovered since the NODE-301 Test Dose Randomization Visit, including those reported on the Cardiac Monitoring System (CMS) report of the outpatient PSVT event treated with the study drug in the NODE 301 study:

   d. Third-degree Atrioventricular (AV) block, Mobitz II second-degree AV block, or Wenckebach with bradycardia ≤40 bpm; e. Significant symptomatic sinus bradycardia heart rate (HR) ≤40 bpm or sinus pauses (≥3 seconds); f. Any significant ventricular arrhythmia (premature ventricular beats and couplets [>6 premature ventricular contractions per 45 seconds electrocardiogram (ECG)] are considered significant); or g. Atrial fibrillation (event lasting longer than 30 seconds);
2. Any drug-related or procedure-related serious adverse event during the NODE-301 study;
3. Any severe adverse event (AE) in the NODE-301 study that was severe enough to preclude administration of etripamil NS 70 mg in the NODE-302 study;
4. Any new drug prescribed after the end of the patient's participation in the NODE-301 study that could lower blood pressure or decrease AV node conduction;
5. Systolic blood pressure <90 mmHg after a 5-minute rest in sitting position at the NODE-302 Qualification Visit;
6. Any symptoms consistent with clinically severe hypotension such as presyncope, medically significant lightheadedness, syncope, nausea, or vomiting;
7. New therapy with digoxin, amiodarone, or any Class I or III antiarrhythmic drug added after the end of the patient's participation in the NODE-301 study;
8. New evidence of ventricular pre-excitation (e.g., delta waves, short PR interval, Wolff Parkinson-White syndrome) on the ECG since randomization in the NODE-301 study;
9. New symptoms of congestive heart failure defined by the New York Heart Association Class II to IV since randomization in the NODE-301 study;
10. New stroke since randomization in the NODE-301 study;
11. New evidence of a significant physical or psychiatric condition including drug abuse, which in the opinion of the Investigator, could jeopardize the safety of the patient, or impede the patient's capacity to follow the study procedures since randomization in the NODE-301 study;
12. New syncope since randomization in the NODE-301 study, especially if observed during the monitoring of the event treated in the NODE-301 study;
13. New evidence of hepatic dysfunction defined as alanine aminotransferase or aspartate aminotransferase >3 × the upper limit of normal (ULN) or total bilirubin >2 × ULN, unless due to Gilbert syndrome observed at the NODE-302 Qualification Visit;
14. New evidence of renal dysfunction as determined by an estimated glomerular filtration rate assessed at the NODE-302 Qualification Visit as follows:

    1. <60 mL/min/1.73 m2 for patients <60 years of age,
    2. <40 mL/min/1.73 m2 for patients ≥60 and <70 years of age, or
    3. <35 mL/min/1.73 m2 for patients ≥70 years of age;
15. Participation in any investigational drug or device study or the use of any investigational drug or device since the Final Study Visit in the NODE-301 study.

Withdrawal Criteria

Patient participation in this clinical study may be discontinued for any of the following reasons:

* The patient withdraws consent or requests discontinuation from the study for any reason;
* The patient took the study drug in both the NODE-301 and the NODE-302 studies for symptoms not associated with an episode of PSVT;
* Occurrence of any medical condition, AE, or circumstance that exposes the patient to substantial risk and/or does not allow the patient to adhere to the requirements of the protocol;
* Requirement of a prohibited concomitant medication and/or change in the use of chronic therapies, such as concomitant beta-blockers, calcium channel blockers, and medications that can lower blood pressure;
* Patient failure to comply with protocol requirements or study-related procedures;
* Termination of the study by Milestone or a regulatory authority; or
* The patient self-administered a total of 11 doses of etripamil Nasal Spray 70 mg in the NODE-302 study.

Patients who withdraw from the study after taking etripamil Nasal Spray 70 mg and had a Follow-up Visit will be required to undergo an Early Termination Visit.

Patients who withdraw from the study and did not take etripamil Nasal Spray 70 mg will be required to undergo an Early Termination Visit.

Patients who withdraw after taking the study drug but did not have a Follow-up Visit will be required to undergo a Final Study Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (22):
  - Arizona Arrhythmia Research Center, Phoenix, Arizona
  - Arkansas Cardiology, Little Rock, Arkansas
  - Los Alamitos Cardiovascular, Los Alamitos, California
  - South Denver Cardiology Associates, P.C, Littleton, Colorado
  - Baptist Health Ambulatory Services, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Edgewater Medical Research, New Smyrna Beach, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Georgia Arrythmia Consultants&Research Institute, Macon, Georgia
  - Iowa Heart Center, West Des Moines, Iowa
  - MedStar Health Research Institute, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Atlantic Health System - Morristown Medical Center, Morristown, New Jersey
  - Trinity Medical WNY, PC, Buffalo, New York
  - Weill Cornell Medical Center, New York, New York
  - The Presbyterian Hospital DBA Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - Heart House Research Foundation, LLC, Springfield, Ohio
  - Black Hills Cardiovascular Research, Rapid City, South Dakota
  - Baylor College of Medicine, Houston, Texas
  - Baylor Scott and White Research Institute - Round Rock, Round Rock, Texas
  - IHC Health Services Inc. DBA Intermountain Medical Center, Murray, Utah
- Canada (12):
  - Libin Cardiovascular Institute of Alberta - University of Calgary, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Vancouver General Hospital - Research Institute ; Gordon and Leslie Diamond Health Centre, Vancouver, British Columbia
  - Victoria Cardiac Arrhythmia Trials, Inc., Victoria, British Columbia
  - University of Manitoba, St Boniface General Hospital, Winnipeg, Manitoba
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Dawson Road Medical Centre, Guelph, Ontario
  - Hamilton Health Sciences, Hamilton, Ontario
  - Partners in Advanced Cardiac Evaluation (PACE) Cardiology Clinic, Newmarket, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Montreal Heart Institute - Institut de Cardiologie de Montréal, Montreal, Quebec
  - CIUSSS de l'Estrie - CHUS ; Hôpital Fleurimont, Sherbrooke, Quebec

REFERENCES:
- [Derived] Ip JE, Coutu B, Bennett MT, Pandey AS, Stambler BS, Sager P, Chen M, Shardonofsky S, Plat F, Camm AJ. Etripamil Nasal Spray for Conversion of Repeated Spontaneous Episodes of Paroxysmal Supraventricular Tachycardia During Long-Term Follow-Up: Results From the NODE-302 Study. J Am Heart Assoc. 2023 Oct 3;12(19):e028227. doi: 10.1161/JAHA.122.028227. Epub 2023 Sep 27. PMID 37753718

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients randomized in Part 1 of the NODE-301 study and who met the inclusion and exclusion criteria of the NODE-302 study were eligible for the NODE-302 study. This study was conducted only at clinical sites that participated in the NODE-301 Part 1 study. Study was initiated on December 10, 2018 and completed on November 13, 2020.
Pre-assignment Details: Of the 169 patients enrolled, 64 (37.9%) of 169 patients did not treat an episode with etripamil in this study.
Groups:
- Etripamil NS 70 mg: The dose of etripamil evaluated in NODE-302 was 70 mg.
  Etripamil NS 70 mg: All patients received a total of 200 micro-liters of etripamil NS 70 mg via the Aptar Pharma Nasal Spray Bidose System each time they self-administer study drug.
  Aptar Pharma Nasal Spray Bidose System: Patients were self-administer the study drug using the Aptar Pharma Nasal Spray Bidose System. The devices were be prefilled and packaged into child-resistant boxes. Instructions for its use was provided in the study drug box.
Period: Overall Study
Arm/Group | Etripamil NS 70 mg
Started | 169
Patients Not Treated With Etripamil | 64
Safety Population | 105
Efficacy Population | 92 (92 patients (from safety population) treated with etripamil for a positively adjudicated episode of PSVT)
Completed | 2 (Early study termination = 167 patients)
Not Completed | 167
Not completed — Study terminated by Sponsor | 94
Not completed — Withdrawal by Subject | 20
Not completed — Ablation | 26
Not completed — Adverse Event | 7
Not completed — Physician Decision | 3
Not completed — Prohibited medication | 5
Not completed — Did not meet eligibility criteria | 5
Not completed — Site closure (2), compliance with IP, directed by sponsor and site termination. | 5
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Safety population
Arm/Group | Etripamil NS 70 mg
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age at informed consent signed | 58 (13.75)
  Age at confirmation of PSVT | 57.2 (13.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 100
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 8
  White | 87
  More than one race | 5
  Unknown or Not Reported | 0
PSVT confirmation duration (years) [Mean (Standard Deviation); unit: years] | 1.3 (1.73)
Number of patient-reported PSVT episodes in the year prior to NODE-301 [Mean (Standard Deviation); unit: episodes] | 9.7 (11.79)
Number of patient-reported emergency department visits for PSVT in lifetime [Mean (Standard Deviation); unit: emergency department visits] — Population: Not all patients reported emergency department visit
  emergency department visits
    number analyzed (Participants) | 103
    (all) | 2.7 (2.74)

OUTCOME MEASURES:

1. Primary Outcome: Time to Conversion of an Episode of PSVT to Sinus Rhythm (SR) After Study Drug Administration.
Description: The efficacy analyses were performed on the Efficacy Population. The primary efficacy variable was the time to conversion of an episode of PSVT to SR after study drug administration.
Time Frame: 18 months
Population: Primary analysis of the primary efficacy endpoint for each patient's first episode of PSVT confirmed by adjudication and treated with etripamil NS 70 mg. There were 92 patients who had a PSVT episode that was confirmed by adjudication and were included in the primary analysis.
Measure: Median (95% Confidence Interval); unit: minutes
Groups:
- Etripamil NS 70 mg: The dose of etripamil evaluated in NODE-302 was 70 mg.
  Etripamil NS 70 mg: All patients received a total of 200 micro-liters of etripamil NS 70 mg via the Aptar Pharma Nasal Spray Bidose System each time they self-administer study drug.
  Aptar Pharma Nasal Spray Bidose System: Patients were self-administer the study drug using the Aptar Pharma Nasal Spray Bidose System. The devices were prefilled and packaged into child-resistant boxes. Instructions for its use was provided in the study drug box.
Arm/Group | Etripamil NS 70 mg
Number analyzed (Participants) | 92
minutes | 21.1 [11.6 to 35.5]

ADVERSE EVENTS:
Time Frame: 18 months.
Description: TEAEs in this study are defined as AEs with a start date occurring 0 to 24 hours after a dose of study drug dose. In the text these are referred to as TEAE24.
Arm/Group | Etripamil NS 70 mg
All-Cause Mortality (participants affected / at risk) | 0/105
Serious Adverse Events (participants affected / at risk) | 8/105
Other Adverse Events (participants affected / at risk) | 67/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etripamil NS 70 mg (N=105)
Bradycardia (Cardiac disorders) | 1 — SAE not related to etripamil
Supraventricular tachycardia (Cardiac disorders) | 3 — SAE not related to etripamil
Ataxia (Nervous system disorders) | 1 — SAE not related to etripamil
Syncope (Nervous system disorders) | 1 — SAE not related to etripamil
Pancreatitis (Gastrointestinal disorders) | 1 — SAE not related to etripamil
Troponin increased (Investigations) | 1 — SAE not related to etripamil
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etripamil NS 70 mg (N=105)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 23
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 17
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Sneezing (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Headache (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 4
Paresthesia (Nervous system disorders) | 2
Mucosal hypertrophy (General disorders) | 5
Lacrimation increased (Eye disorders) | 3
Heart rate increased (Investigations) | 3
Atrial fibrillation (Cardiac disorders) | 3
Eye irritation (Eye disorders) | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 4
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 3
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Increased viscosity of upper respiratory secretion (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/96/NCT03635996/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT03635996/SAP_001.pdf